CLINICAL TRIAL: NCT06702982
Title: Virtual Support, Real Impact: the Effectiveness of Tele-nursing in Alleviating Chemotherapy Symptoms Among Cancer Patients; a Quasi-experimental Study
Brief Title: Virtual Support, Real Impact: Effectiveness of Tele-nursing in Alleviating Chemotherapy Symptoms Among Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Alaa El Din Moustafa Hamed Abd Elaleem, Lecturer of Psychiatric and mental health Nursing, Helwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NURRSC23071035
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Chemotherapy Effect; Quality of Life (QOL)
Keywords: chemotherpay; tele-nursing; quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enrolled participants (Experimental): The intervention administered in this study was a tele-nursing educational program aimed at improving cancer patients' management of chemotherapy-related symptoms and enhancing their quality of life. The program was delivered via a Telegram group, which provided a platform for regular interaction between the patients and nursing staff. The educational content was designed to address common chemotherapy-related symptoms, such as nausea, fatigue, pain, and loss of appetite, and to provide guidance on managing these symptoms effectively.
  Interventions: Behavioral: tele-nursing educational program

INTERVENTIONS:
Behavioral: tele-nursing educational program — The intervention administered in this study was a tele-nursing educational program aimed at improving cancer patients' management of chemotherapy-related symptoms and enhancing their quality of life. The program was delivered via a Telegram group, which provided a platform for regular interaction between the patients and nursing staff. The educational content was designed to address common chemotherapy-related symptoms, such as nausea, fatigue, pain, and loss of appetite, and to provide guidance on managing these symptoms effectively.

SUMMARY:
This quasi-experimental study evaluated a tele-nursing educational program's impact on improving the quality of life and managing chemotherapy-related symptoms in 74 adult cancer patients at Mansoura University Hospital in Egypt. Delivered via Telegram, the program involved weekly educational sessions, aiming to enhance symptom management and quality of life.

DETAILED DESCRIPTION:
The study aimed to assess the effectiveness of a tele-nursing educational program in managing chemotherapy-related and cancer-related symptoms and improving the quality of life among adult cancer patients. Conducted at the Oncology Center at Mansoura University Hospital in Egypt, the study recruited 74 participants who completed structured interviews detailing their demographics, medical history, symptom severity (using the MDASI-A tool), and quality of life (using the QOL-ACD tool). The intervention, delivered via a Telegram group, included weekly educational sessions focused on managing chemotherapy symptoms. The sessions featured educational content and feedback, with outcomes measured through changes in symptom severity and quality of life scores before and after the intervention. This approach highlighted the program's potential to enhance patients' overall well-being and symptom management.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with cancer and receiving treatment at an outpatient chemotherapy center

  * Age from 20 less than 60 years.
  * Accept to participate in the study.
  * Had smart phones linked with internet
  * Educated and able to use Zoom and Telegram applications

Exclusion Criteria:

* • Having active, serious physical disease

  * Patients with mental disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
cancer-related and treatment-related symptoms | 3 months
  The M.D. Anderson Symptom Inventory Arabic Version (MDASI-A), adapted from Nejmi et al. (2010), was utilized to assess the severity of cancer-related and treatment-related symptoms in a manner accessible to Arabic-speaking patients. Designed in straightforward Arabic, the tool evaluates both the intensity of 13 core symptoms commonly experienced by cancer patients and their interference with daily functioning. This makes the MDASI-A comprehensive while remaining brief enough to avoid imposing a burden on respondents.
  The MDASI-A employs a 0-2 numerical scale (Never = 0, Sometimes = 1, Always = 2), ensuring its usability even among less-educated individuals. It is also adaptable for telephone, computer, and other electronic methods of administration. Scores were converted to percentages to classify symptom intensity into three categories: low (<50%), average (50% to <75%), and high (≥75%) based on the method proposed by Daisuke and Makoto (2022).

SECONDARY OUTCOMES:
Quality of life for Cancer Patients | 3 months
  The Quality of Life Questionnaire for Cancer Patients Treated with Anticancer Drugs (QOL-ACD), adopted from Kurihara et al. (1999), was employed to assess the quality of life (QOL) among patients undergoing anticancer treatment. This questionnaire comprises 22 items distributed across five domains: six items for daily activities, five for physical condition, five for mental and psychological status, five for social activities, and one for general QOL (evaluated via a face scale). Each item was rated on a 5-point scale, with scores ranging from 1 (lowest QOL) to 5 (highest QOL), yielding a total score between 22 and 110; higher scores indicate better QOL.
  Patients' responses were classified into three categories based on their scores: good (≤75%), average (50%-<75%), and low (>50%), according to the scoring framework by Saad and Elsayed (2021). Negative statements were reverse scored to align with the Likert scale format, ensuring consistency in the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El Din M Abd Elaleem, PhD, Principal Investigator — Faculty of Nursing
Locations (1):
- Mansura university, Al Mansurah, Dakhalia, Egypt

IPD SHARING:
Plan to Share IPD: No